CLINICAL TRIAL: NCT00090857
Title: A Pilot Study of Aromatase Inhibitors for Women at Increased Risk of Breast Cancer Based on Estradiol Levels
Brief Title: Letrozole in Preventing Breast Cancer in Postmenopausal Women
Acronym: WISE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Jonsson Comprehensive Cancer Center (Other)
Responsible Party: Principal Investigator, Judy E. Garber, MD, Garber, Judith MD, Dana-Farber Cancer Institute
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: DFCI-00024; P50CA089393 (NIH); P30CA006516 (NIH); DFCI-00024; UCLA-0210012-02; NCT00165529 (obsolete NCT alias); NCT00577551 (obsolete NCT alias)
Record Dates: First submitted 2004-09-07; First posted 2004-09-08 (Estimated); Results first posted 2017-06-29 (Actual); Last update posted 2018-03-30 (Actual); Status verified 2018-03

CONDITIONS: Breast Cancer
Keywords: breast cancer; stage I breast cancer; stage II breast cancer; stage IIIA breast cancer; stage IIIB breast cancer; stage IIIC breast cancer; stage IV breast cancer; breast cancer in situ; ductal breast carcinoma in situ
MeSH Terms: conditions — Breast Neoplasms; Breast Carcinoma In Situ; Carcinoma, Intraductal, Noninfiltrating | interventions — Letrozole

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Letrozole (Experimental): Participants in this arm received 2.5 mg of letrozole per day for a duration of 12 months; followed by an optional 4 years. Treatment continued in the absence of unacceptable toxicity or diagnosis of invasive breast cancer, ductal carcinoma in situ, or any non-breast primary cancer.
  Interventions: Drug: Letrozole
- Placebo (Placebo Comparator): Participants in this arm received 1 tablet per day which contained the inert ingredients from the letrozole tablet, for a duration of 12 months; followed by an optional 5 years of letrozole.Treatment continued in the absence of unacceptable toxicity or diagnosis of invasive breast cancer, ductal carcinoma in situ, or any non-breast primary cancer.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Letrozole
  Other Names: Femara
  Arms: Letrozole
Other: Placebo
  Arms: Placebo

SUMMARY:
RATIONALE: Chemoprevention therapy is the use of certain drugs to try to prevent the development or recurrence of cancer. Letrozole may be effective in preventing the development or recurrence of breast cancer in postmenopausal women who are at increased risk of developing breast cancer because of elevated estradiol levels.

PURPOSE: This randomized phase II trial is studying how well letrozole works in preventing breast cancer in postmenopausal women with elevated estradiol levels.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* The primary outcome of the study is the change in bone mineral density following a year on letrozole vs. a year on placebo.

Secondary

* Compare the safety, acceptability, and adherence to letrozole vs placebo in postmenopausal women at increased risk for the development or recurrence of breast cancer based on elevated plasma estradiol levels through evaluation of menopausal symptoms (including hot flushes, weight changes, sexual functioning, and genitourinary effects), blood lipid levels, markers of bone turnover, and multidimensional quality of life.
* Determine the effect of letrozole-induced reduction of plasma estradiol levels on mammographic percent breast density.
* Obtain background information for a future large chemoprevention trial to address the question of whether a reduction in plasma estradiol levels can reduce the risk of breast cancer in postmenopausal women.

OUTLINE: This is a pilot, randomized, double-blind, placebo-controlled, multicenter study. Patients are randomized to 2:1 (experimental treatment: placebo arms).

PROJECTED ACCRUAL: A total of 110 patients (73 for arm I and 37 for arm II) will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* At increased risk for the development or recurrence of breast cancer, defined as an estradiol level ≥ 9 pg/mL
* No evidence of suspicious or malignant disease, based on the following examinations:

  * Clinical bilateral breast examination within the past 6 months
  * Bilateral* mammogram within 3 months before randomization OR within 30 days after randomization
  * Pelvic exam normal within the past 5 years
  * General physical exam within the past 6 months NOTE: *Unilateral mammogram of the uninvolved breast for patients with prior invasive breast cancer or ductal carcinoma in situ (DCIS)
* Bone density scan within 2 standard deviations from normal within the past 30 days

  * Bone density scan ≥ 2 standard deviations below normal allowed if approved by the study physician
* At least 1 breast that has not been previously treated with radiotherapy or surgery (for patients with prior invasive breast cancer or DCIS)
* Hormone receptor status:

  * Not specified

PATIENT CHARACTERISTICS:

Age

* 35 and over

Sex

* Female

Menopausal status

* Postmenopausal, defined by any of the following criteria:

  * At least 12 months without spontaneous menstrual bleeding
  * Prior hysterectomy and bilateral salpingo-oophorectomy
  * ≥ 55 years of age with a prior hysterectomy with or without oophorectomy
  * < 55 years of age with a prior hysterectomy without oophorectomy OR the status of the ovaries is unknown AND follicle-stimulating hormone (FSH) level is in the postmenopausal range

Performance status

* Normal activity must not be restricted for a significant portion of the day

Life expectancy

* At least 10 years

Hematopoietic

* Complete blood count with differential normal

  * Prior benign neutropenia allowed provided the granulocyte count is ≥ 1,500/mm^3

Hepatic

* Bilirubin normal
* Alkaline phosphatase normal
* SGOT and SGPT normal

Renal

* Creatinine normal

Cardiovascular

* No uncontrolled cardiovascular disease

Other

* Not pregnant
* No other malignancy within the past 5 years except basal cell or squamous cell skin cancer or carcinoma in situ of the cervix
* No osteoporosis
* No hyperlipidemia
* No mental health status resulting in cognitive or emotional impairment that would preclude study participation

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* Not specified

Endocrine therapy

* More than 30 days since prior AND no concurrent use of any of the following hormonal agents:

  * Estrogen or progesterone replacement therapy
  * Oral contraceptives
  * Raloxifene or other plasma estrogen receptor modulators (SERMs)
  * Androgens (e.g., danazol)
  * Luteinizing hormone-releasing hormone (LHRH) analogs (e.g., goserelin or leuprolide)
  * Prolactin inhibitors (e.g., bromocriptine)
  * Antiandrogens (e.g., cyproterone)
* More than 60 days since prior AND no concurrent tamoxifen
* No prior aromatase inhibitors (for patients with prior invasive breast cancer or DCIS)
* No concurrent phytoestrogenic dietary supplements (e.g., soy, ginseng, or other natural products)

  * Dietary soy allowed

Radiotherapy

* See Disease Characteristics

Surgery

* See Disease Characteristics
* No prior bilateral mastectomy

Other

* More than 60 days since prior treatment for invasive breast cancer or DCIS
* More than 30 days since prior bisphosphonates or calcitonin
* No prior or concurrent participation on a treatment study for invasive breast cancer or DCIS
* No concurrent participation in any other cancer prevention study or osteoporosis prevention study involving pharmacologic agents
* No concurrent calcitonin
* No concurrent bisphosphonate therapy
* Concurrent cholecalciferol (vitamin D) and calcium to augment bone mineral density allowed

Ages: 35 Years to 120 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2002-02 (Actual); Primary Completion 2008-08 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Judy Garber, MD, Principal Investigator — Dana-Farber Cancer Institute; Patricia A. Ganz, MD, Principal Investigator — Jonsson Comprehensive Cancer Center
Locations (5):
- United States (5):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana-Farber/Harvard Cancer Center at Dana Farber Cancer Institute, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Dan L. Duncan Cancer Center at Baylor College of Medicine, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients enrolled from February 2002 through August 2007.
Pre-assignment Details: In this chemoprevention trial, postmenopausal women were screened and eligible based on serum estradiol levels. Of 405 women screened, 381 were eligible for blood draw. Of these 381 women eligible for blood draw, 87 were eligible for randomization based on serum estradiol level (>/=0.9 ng/dL). There were 38 women who declined to be randomized.
Period: Overall Study
Arm/Group | Letrozole | Placebo
Started | 33 | 16
Completed | 29 | 13
Not Completed | 4 | 3
Not completed — Lost to Follow-up | 0 | 1
Not completed — Withdrawal by Subject | 2 | 0
Not completed — Adverse Event | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Letrozole | Placebo | Total
Number analyzed (Participants) | 33 | 16 | 49
Age, Continuous [Median (Full Range); unit: years] | 56 [45 to 66] | 52.5 [48 to 72] | 54 [45 to 72]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33 | 16 | 49
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 33 | 16 | 49

OUTCOME MEASURES:

1. Primary Outcome: Change in Lumbar Density From Baseline to 12 Months
Description: The bone mineral density (BMD) test was comprised of the following 4 measurements [total density (g/cm^2)]: lumbar, femoral neck, trochanter, hip.
Time Frame: Evaluation occurred at treatment initiation (BL) and after 12-months of treatment.
Population: The analysis dataset is comprised of randomized patients with an evaluable sample for analysis of lumbar density.
Measure: Median (Full Range); unit: g/cm^2
Arm/Group | Letrozole | Placebo
Number analyzed (Participants) | 29 | 13
g/cm^2 | -0.036 [-0.092 to 0.272] | -0.021 [-0.180 to 0.064]
Statistical Analysis 1: Comparison: Letrozole vs Placebo; Sample size for a detectable difference in the within participant change in bone density between arms was calculated using standard deviations of one year change in bone density. Control estimates were 2.8% for spine and 3.85% for femoral neck. With 100 patients and 2:1 randomization (67 letrozole: 33 placebo), using a 1-sided Wilcoxon rank sum test with size 0.05, there is 80% power to detect as significant a true difference in change in the spine of 1.6% and in the femoral neck of 2.27%; Test type: Superiority or Other; p = 0.15, Wilcoxon (Mann-Whitney)

2. Primary Outcome: Change in Femoral Neck Density From Baseline to 12 Months
Description: as for outcome 1
Time Frame: Evaluation occurred at treatment initiation (BL) and after 12-months of treatment.
Population: The analysis dataset is comprised of randomized patients with an evaluable sample for analysis of femoral neck density.
Measure: Median (Full Range); unit: g/cm^2
Arm/Group | Letrozole | Placebo
Number analyzed (Participants) | 28 | 13
g/cm^2 | -0.0065 [-0.097 to 0.068] | -0.013 [-0.13 to 0.029]
Statistical Analysis 1: Comparison: Letrozole vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.70, Wilcoxon (Mann-Whitney)

3. Primary Outcome: Change in Trochanter Density From Baseline to 12 Months
Description: as for outcome 1
Time Frame: Evaluation occurred at treatment initiation (BL) and after 12-months of treatment.
Population: The analysis dataset is comprised of randomized patients with an evaluable sample for analysis of trochanter density.
Measure: Median (Full Range); unit: g/cm^2
Arm/Group | Letrozole | Placebo
Number analyzed (Participants) | 27 | 13
g/cm^2 | -0.017 [-0.059 to 0.023] | -0.009 [-0.059 to 0.015]
Statistical Analysis 1: Comparison: Letrozole vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.03, Wilcoxon (Mann-Whitney)

4. Primary Outcome: Change in Hip Density From Baseline to 12 Months
Description: as for outcome 1
Time Frame: Evaluation occurred at treatment initiation (BL) and after 12-months of treatment.
Population: The analysis dataset is comprised of randomized patients with an evaluable sample for analysis of hip density.
Measure: Median (Full Range); unit: g/cm^2
Arm/Group | Letrozole | Placebo
Number analyzed (Participants) | 28 | 13
g/cm^2 | -0.0275 [-0.082 to 0.035] | -0.001 [-0.075 to 0.025]
Statistical Analysis 1: Comparison: Letrozole vs Placebo; Sample size for a detectable difference in the within participant change in bone density was calculated using standard deviations of one year change in bone density. Control estimates were 2.8% for spine and 3.85% for femoral neck. With 100 patients and 2:1 randomization (67 letrozole: 33 placebo), using a 1-sided Wilcoxon rank sum test with size 0.05, there is 80% power to detect as significant a true difference in change in the spine of 1.6% and in the femoral neck of 2.27%; Test type: Superiority or Other; p = 0.06, Wilcoxon (Mann-Whitney)

5. Secondary Outcome: Worst Grade Hot Flashes
Description: Participants reported worst grade hot flashes: 01: mild (<1qd) or 02: moderate (>1qd) during 12 months of treatment.
Time Frame: Heath assessments during treatment were administered at 3- and 9-months by telephone contact and during clinic visits at 6- and12-months.
Population: The analysis dataset is comprised of all randomized participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Letrozole | Placebo
Number analyzed (Participants) | 33 | 16
Participants
  None | 14 | 9
  Mild (<1 qd) | 5 | 3
  Moderate | 11 | 4
  Missing | 3 | 0
Statistical Analysis 1: Comparison: Letrozole vs Placebo; Test type: Superiority or Other; p = 0.38, Fisher Exact

6. Secondary Outcome: Worst Grade Muscle Aches/Pains
Description: Participants reported worst grade muscle aches/pains defined as grade 01: mild, 02: moderate, 03: severe (CTCAEv3) or 04: disabling (CTCAEv3) during 12 months of treatment.
Time Frame: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Letrozole | Placebo
Number analyzed (Participants) | 33 | 18
Participants
  None | 14 | 13
  Mild | 8 | 2
  Moderate | 7 | 1
  Severe | 1 | 0
  Missing | 3 | 0
Statistical Analysis 1: Comparison: Letrozole vs Placebo; Test type: Superiority or Other; p = 0.02, Fisher Exact

7. Secondary Outcome: Worst Grade Nausea
Description: Participants reported worst grade nausea grade 01: able to eat, 02: oral intake significantly decreased, 03: no significant intake, requiring IV fluids during 12 months of treatment.
Time Frame: as for outcome 5
Population: The analysis dataset is comprised of all randomized participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Letrozole | Placebo
Number analyzed (Participants) | 33 | 16
Participants
  None | 23 | 15
  Able to Eat | 5 | 1
  Oral Intake Significantly Decreased | 1 | 0
  Missing | 4 | 0
Statistical Analysis 1: Comparison: Letrozole vs Placebo; Test type: Superiority or Other; p = 0.20, Fisher Exact

8. Secondary Outcome: Worst Grade Vomiting
Description: Participants reported worst grade vomiting grade 01: 1x in 24 hours, 02: 2-5x in 24 hours, 03: >/= 6x in 24 hours, grade 04: requiring parenteral nutrition/intensive care during 12 months of treatment.
Time Frame: as for outcome 5
Population: The analysis dataset is comprised of all randomized participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Letrozole | Placebo
Number analyzed (Participants) | 33 | 16
Participants
  None | 28 | 15
  1x in 24 hours | 1 | 0
  2-5x in 24 hours | 0 | 1
  Missing | 4 | 0
Statistical Analysis 1: Comparison: Letrozole vs Placebo; Test type: Superiority or Other; p = .88, Fisher Exact

9. Secondary Outcome: Worst Grade Abdominal Pain
Description: Participants reported worst grade abdominal pain: 01: mild, 02: moderate, 03: severe (CTCAEv3), 04: disabling (CTCAEv3) during 12 months of treatment.
Time Frame: as for outcome 5
Population: The analysis dataset is comprised of all randomized participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Letrozole | Placebo
Number analyzed (Participants) | 33 | 16
Participants
  None | 27 | 16
  Mild | 3 | 0
  Missing | 3 | 0
Statistical Analysis 1: Comparison: Letrozole vs Placebo; Test type: Superiority or Other; p = 0.27, Fisher Exact

10. Secondary Outcome: Worst Grade Bone Pain
Description: Participants reported worst grade bone pain: 01: mild, 02: moderate, 03: severe (CTCAEv3), 04: disabling (CTCAEv3) during 12 months of treatment.
Time Frame: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Letrozole | Placebo
Number analyzed (Participants) | 33 | 16
Participants
  None | 22 | 12
  Mild | 2 | 3
  Moderate | 6 | 1
  Missing | 3 | 0
Statistical Analysis 1: Comparison: Letrozole vs Placebo; Test type: Superiority or Other; p = .60, Fisher Exact

11. Secondary Outcome: Worst Grade Headache
Description: Participants reported worst grade headache: 01: mild, 02: moderate, 03: severe (CTCAEv3), 04: disabling (CTCAEv3) during 12 months of treatment.
Time Frame: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Letrozole | Placebo
Number analyzed (Participants) | 33 | 16
Participants
  None | 20 | 11
  Mild | 7 | 3
  Moderate | 3 | 2
  Missing | 3 | 0
Statistical Analysis 1: Comparison: Letrozole; Test type: Superiority or Other; p = .58, Fisher Exact

12. Secondary Outcome: Worst Grade Fatigue
Description: Participants reported worst grade fatigue: 01: mild, 02: moderate, 03: severe (CTCAEv3), 04: disabling (CTCAEv3) during 12 months of treatment.
Time Frame: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Letrozole | Placebo
Number analyzed (Participants) | 33 | 16
Participants
  None | 19 | 11
  Mild | 6 | 2
  Moderate | 5 | 3
  Missing | 3 | 0
Statistical Analysis 1: Comparison: Letrozole vs Placebo; Test type: Superiority or Other; p = .49, Fisher Exact

ADVERSE EVENTS:
Time Frame: Adverse events were evaluated and reported on the case report forms while participants were on randomized treatment at each clinic follow-up visit (months 6 and 12). If participants opted to continue treatment beyond 12 months then adverse events were monitored annually. Relevant for this report were the adverse events associated with the planned 12 months of treatment. 86% of patients in this study cohort completed 12 months of randomized treatment (median treatment duration is 12 months).
Description: Serious adverse events (SAEs) per protocol were defined as follows: 1) death, 2) a life-threatening adverse drug experience, 3) inpatient hospitalization or prolongation of existing hospitalization, 4) a persistent or significant disability/incapacity, or 5) a congenital anomaly/birth defect. All remaining AEs are Other AEs. Of note, secondary outcome measures 5-12 provide data on pre-specified analyses of key symptoms pertaining to use of the experimental treatment.
Groups:
- Placebo: Participants in this arm received 1 tablet per day which contained the inert ingredients from the letrozole tablet, for a duration of 12 months; followed by an optional 5 years of letrozole. Treatment continued in the absence of unacceptable toxicity or diagnosis of invasive breast cancer, ductal carcinoma in situ, or any non-breast primary cancer.
Arm/Group | Letrozole | Placebo
All-Cause Mortality (participants affected / at risk) | 0/33 | 0/16
Serious Adverse Events (participants affected / at risk) | 1/33 | 0/16
Other Adverse Events (participants affected / at risk) | 6/33 | 2/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Letrozole (N=33) | Placebo (N=16)
Pain - Head/Headache (Nervous system disorders) | 1 (1) | 0 (0)
Urticaria (hives, welts, wheals) (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Pruritus / Itching (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Letrozole (N=33) | Placebo (N=16)
Arthritis (non-septic) (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain - Muscle (Musculoskeletal and connective tissue disorders) | 2 | 1
Vaginitis (not due to infection) (Reproductive system and breast disorders) | 1 | 0
Vasovagal episode (Nervous system disorders) | 0 | 1
Dizziness (Nervous system disorders) | 1 | 0
Weight gain (Investigations) | 1 | 0
Fatigue (asthenia, lethargy, malaise) (General disorders) | 1 | 0
Hot flashes/flushes (Vascular disorders) | 1 | 0
Pain - Chest/thorax NOS (General disorders) | 1 | 0
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 1 | 0

LIMITATIONS AND CAVEATS:
Results on this study are limited due to the age of the trial and the prior departure of the coordinator who assisted with the data collection. The accrual goal was not met with many participants eligible upon screening declining randomization.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No